CLINICAL TRIAL: NCT06769217
Title: A Prospective Multi-Centre Registry of EvroSure (Everolimus Drug Eluting CoCr Coronary Stent)to Investigate Safety and Effectiveness Nam of Study:EverGreen
Brief Title: Clinical Investigation for Everolimus Drug Eluting Stent
Acronym: EverGreen
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Frisch Medical Device Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESC/FM/030622
Record Dates: First submitted 2025-01-03; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: A Prospective Multi-Centre Registry for Everolimus Drug Eluting CoCr Coronary Stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other): Its a single arm multicenter registry to investigate safety and efficacy of product by clinical follow up at one month and 12 month
  Interventions: Device: Drug Eluting Coronary Stent

INTERVENTIONS:
Device: Drug Eluting Coronary Stent — The Drug Eluting Coronary stent is indicated for the treatment of de novo coronary artery lesions in patients with symptomatic ischemic heart disease.

SUMMARY:
History of Device Development and Study Rationale:

Drug-eluting stents (DES) revolutionized percutaneous coronary intervention (PCI) by significantly reducing restenosis and the need for repeat procedures compared to bare-metal stents (BMS). Introduced in the early 2000s, DES quickly became the standard of care due to its superior antiproliferative properties.

DES consist of a metal stent, an antiproliferative drug, and a polymer coating. The stent provides structural support while the drug is gradually released to inhibit tissue growth within the artery. This dual action effectively prevents restenosis, a common complication after PCI.

Contemporary guidelines strongly recommend DES over BMS for various clinical scenarios. The proven efficacy and safety of current-generation DES make them the preferred treatment option for patients undergoing PCI.

First-generation drug-eluting stents:

First-generation drug-eluting stents (DES) marked a significant advancement in interventional cardiology, addressing the persistent issue of in-stent restenosis (ISR) associated with bare-metal stents (BMS). These innovative devices, composed of a metal frame, an antiproliferative drug (sirolimus or paclitaxel), and a polymer coating, were designed to release the drug gradually, preventing tissue growth within the artery. Clinical trials demonstrated the superior efficacy of DES over BMS in reducing ISR and target lesion revascularization (TLR). The RAVEL trial, for example, found a dramatic decrease in ISR with sirolimus-eluting stents (SES). Subsequent studies and meta-analyses confirmed the benefits of both SES and paclitaxel-eluting stents (PES) compared to BMS, particularly in high-risk patients.

The introduction of DES represented a paradigm shift in interventional cardiology, offering a more effective and durable solution for patients with coronary artery disease.

Second-generation drug-eluting stents:

Second-generation drug-eluting stents (DES) were developed to address the safety concerns associated with first-generation DES, such as stent thrombosis (ST), incomplete endothelialisation, and polymer-induced inflammation. These newer stents incorporate less toxic drugs, more biocompatible coatings, and thinner, more flexible struts. Clinical trials have demonstrated the superior safety and efficacy of second-generation DES compared to their predecessors. Studies comparing everolimus-eluting stents (EES) and zotarolimus-eluting stents (ZES) to first-generation DES have shown significant reductions in ST, myocardial infarction (MI), and target lesion revascularisation (TLR). Head-to-head comparisons of EES and ZES have also revealed comparable outcomes in real-world patient populations. Both stents are effective and safe for the treatment of obstructive coronary artery disease, making them the preferred choice for percutaneous coronary intervention.

Study Rationale:

The introduction of drug-eluting stents (DES) marked a significant leap in interventional cardiology by addressing the limitations of bare-metal stents (BMS), primarily through reducing restenosis and the need for repeat procedures. First-generation DES, equipped with antiproliferative drugs like sirolimus and paclitaxel, demonstrated superior efficacy in preventing in-stent restenosis. However, safety concerns, including stent thrombosis and polymer-induced inflammation, led to the development of second-generation DES, which utilises more biocompatible materials and refined designs. Clinical trials have consistently shown that these newer DES offer enhanced safety and effectiveness, solidifying their position as the preferred treatment option in percutaneous coronary interventions.

Study Objectives

The main objective of this study is to assess the safety and effectiveness of the EvroSure Everolimus Drug eluting CoCr stent in obstructive coronary artery disease.

Primary Objective

The primary endpoint of this study is to monitor Major Adverse Cardiac Events (MACE) at 30 days.

Secondary Objective

The following secondary effectiveness endpoints are as follows:

* Angiographic/device success (%)
* Procedural success (%)
* Clinically justified Target Lesion Revascularization (TLR) (%) at 12 months

The following secondary safety endpoints are:

* MACE (%) until 12 months (Clinically Justified)
* Device-related SAEs until 12 months (Clinically Justified)

Note: MACE rate is defined as the incidence of the combined clinical endpoint: Composite of Death (Cardiac death as well as Non-Cardiac), Myocardial Infarction (Q-wave and non-Q-wave), Emergency Coronary Artery Bypass Graft Surgery, clinically justified TLR following index procedure.

DETAILED DESCRIPTION:
10. Study Objectives The main objective of this study is to assess the safety and effectiveness of the EvroSure Everolimus Drug eluting CoCr stent in obstructive coronary artery disease.

Primary Objective The primary endpoint of this study is to monitor Major Adverse Cardiac Events (MACE) at 30 days.

Secondary Objective

The following secondary effectiveness endpoints are as follows:

* Angiographic/device success (%)
* Procedural success (%)
* Clinically justified Target Lesion Revascularization (TLR) (%) at 12 months

The following secondary safety endpoints are:

* MACE (%) until 12 months (Clinically Justified)
* Device-related SAEs until 12 months (Clinically Justified) Note: MACE rate is defined as the incidence of the combined clinical endpoint: Composite of Death (Cardiac death as well as Non-Cardiac), Myocardial Infarction (Q-wave and non-Q-wave), Emergency Coronary Artery Bypass Graft Surgery, clinically justified TLR following index procedure.

Study Endpoints

Primary endpoints

The primary endpoint of the study is defined as Major Adverse Cardiac Events (MACE) at 30 days.

Note: MACE rate is defined as the incidence of the combined clinical endpoint: Composite of Death (Cardiac death as well as Non-Cardiac), Myocardial Infarction (Q-wave and non-Q-wave), Emergency Coronary Artery Bypass Graft Surgery, clinically justified TLR within 30 days following index procedure.

Secondary endpoints

The secondary effectiveness endpoints were as follows:

* Angiographic/device success (%) (Angiographic device success is determined by confirming the accurate placement of the device within the targeted coronary arteries through X-ray examination.)
* Procedural success (%) (Procedural success is determined by successful implantation of the stent and clearance of blockage.)
* Clinically justified Target Lesion Revascularization (TLR) (%) at 12 months

The following secondary safety endpoints were assessed:

* MACE (%) until 12 months (Clinically Justified)
* Device-related SAEs until 12 months (Clinically Justified)

ELIGIBILITY:
Inclusion Criteria:

-1. The patient must be ≥ 18 years of age; 2. Patient was an acceptable candidate for PTCA, Stenting, or Emergent CABG; 3. Patient has clinical evidence of ischemic heart disease or a positive functional study 4. Patient and his or her treating physician agree that the patient will comply with all the required post-procedure follow-up.

5. Target lesion(s) present with ≥50% stenosis, in one or more vessels 6. Target lesions have to be de novo; 7. One or more target lesions require treatment 8. Reference vessel diameter of target lesion(s) must be ≥ 2.25mm and ≤ 4.5mm, by visual estimate

Exclusion Criteria:

* 1. Previous PTCA with any stent 2. History of CVA or TIA within the last 3 months 3. Patient has active infection 4. Concurrent medical condition with a life expectancy of less than 12 months 5. Clinically relevant contraindication to aspirin, heparin, clopidogrel bisulphate, or ticlopidine including thrombocytopenia, neutropenia, or leukopenia 6. Active peptic ulcer or upper gastrointestinal bleeding. 7. Current participation in an investigational drug or device trial that has not completed its primary endpoint follow-up period.

  8. Pregnancy or woman of childbearing potential who, in the opinion of the investigator, does not take adequate measures to prevent conception.

  9. Known hypersensitivity or contraindication to cobalt, chromium, or nickel

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 888 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is defined as Major Adverse Cardiac Events (MACE) at 30 days. | 30 days
  The primary endpoint of the study is defined as Major Adverse Cardiac Events (MACE) at 30 days.
  Note: MACE rate is defined as the incidence of the combined clinical endpoint: Composite of Death (Cardiac death as well as Non-Cardiac), Myocardial Infarction (Q-wave and non-Q-wave), Emergency Coronary Artery Bypass Graft Surgery, clinically justified TLR within 30 days following index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavin Oza, Bsc, Study Chair — Frisch Medical Devices
Locations (3):
- Baroda Heart Institute & Research Centre, Vadodara, Gujarat, India
- Indonesia (2):
  - Grandmed Lubuk Pakam Hospita, Tanjung Morawa, North Sumatra
  - Primaya Tangerang, Jakarta

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Results
Supporting Information: Study Protocol, CSR
Time Frame: IPD can be shared from 30th January 2025 till 29th January 2026
Access Criteria: Any cardiologist, researcher or author of reputed journals will be able to access, protocol and CER. SomeOne who needs access has to email to frischmedical@gmail.com